CLINICAL TRIAL: NCT02527083
Title: Influence of Anesthetic Technique on Acute and Chronic Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO00000878
Record Dates: First submitted 2015-01-27; First posted 2015-08-18 (Estimated); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2021-05

CONDITIONS: Acute Pain; Chronic Pain; Hernia; Anesthesia, Intravenous; Anesthesia, Intratracheal
MeSH Terms: conditions — Acute Pain; Chronic Pain; Hernia | interventions — Propofol; Sevoflurane; Remifentanil; Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- BIA (Active Comparator): Balanced Inhalational Anesthesia (consisting of a sevoflurane inhaled anesthestic only)
  Interventions: Drug: Sevoflurane; Drug: Remifentanil
- TIVA-K (Active Comparator): Total intravenous anesthetic with ketamine
  Interventions: Drug: Propofol; Drug: Ketamine
- TIVA-R (Active Comparator): Total intravenous anesthetic with remifentanil
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Propofol
  Other Names: Diprivan
  Arms: TIVA-K; TIVA-R
Drug: Sevoflurane
  Other Names: Ultane
  Arms: BIA
Drug: Remifentanil
  Other Names: Ultiva
  Arms: BIA; TIVA-R
Drug: Ketamine
  Other Names: Ketalar
  Arms: TIVA-K

SUMMARY:
Research suggests that the type of anesthesia used for surgery may affect intraoperative stress hormone levels. There is also data to support that an increased level of stress hormones leads to increased pain after surgery. The primary aim of this study is to determine the effect of anesthesia type on long term pain after hernia surgery. In this study, patients undergoing inguinal hernia repair will be randomized to an anesthetic group, either Total Intravenous Anesthesia (TIVA) maintained with propofol or Balanced Inhaled Anesthesia (BIA) maintained with sevoflurane. This will allow us to look at any differences in short and long-term pain after hernia repair depending on type of anesthesia received.

ELIGIBILITY:
Inclusion Criteria:

* All male patients undergoing herniorrhaphy surgery that requires general anesthesia.

Exclusion Criteria:

* Subjects unable to communicate directly with the investigators, due to being non-English speaking, loss of hearing, or incompetence.
* A history of malignant hyperthermia, pseudocholinesterase deficiency, or other disease that prevents anesthetic randomization.
* Pain-related disorders such as fibromyalgia or other chronic pain syndromes.
* Emergency surgery.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- BALANCED INHALATIONAL: Balanced Inhalational Anesthesia (consisting of a sevoflurane inhaled anesthestic only)
  Sevoflurane
  Remifentanil
- TIVA-K: Total intravenous anesthetic with ketamine
  Propofol
  Ketamine
- TIVA-R: Total intravenous anesthetic with remifentanil
  Propofol
  Remifentanil
Period: Overall Study
Arm/Group | BALANCED INHALATIONAL | TIVA-K | TIVA-R
Started | 6 | 2 | 2
Completed | 6 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BALANCED INHALATIONAL | TIVA-K | TIVA-R | Total
Number analyzed (Participants) | 6 | 2 | 2 | 10
Age, Continuous [Mean (Full Range); unit: years] | 65.5 [61 to 69] | 68 [68 to 68] | 73 [68 to 78] | 67.5 [61 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 2 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 2 | 2 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 2 | 10
Pain level in PACU [Mean (Standard Deviation); unit: Pain score (0-10)] — Pain as measured by the Intensity Score of the Pain Quality Assessment Scale (PQAS) in the Post Anesthesia Recovery Unit (PACU) immediately after surgery. The scale goes from 0 (no pain) to 10 (the most intense pain sensation imaginable).
  Pain score (0-10) | 6 (2.68) | 6.5 (4.95) | 6.5 (3.54) | 6.2 (2.86)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score, Chronic
Description: Pain as measured by the Intensity Score of the Pain Quality Assessment Scale (PQAS) at each of the time points after surgery. The scale goes from 0 (no pain) to 10 (the most intense pain sensation imaginable). Higher scores mean worse pain.
Time Frame: 1 month, 3 months, 6 months, 12 months
Population: Only 10 subjects were enrolled, and the numbers represented a typical distribution of Inhalational to TIVA use. Because of the low subject numbers, statistical differences between the techniques were not sought.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BALANCED INHALATIONAL | TIVA-K | TIVA-R
Number analyzed (Participants) | 6 | 2 | 2
score on a scale
  1 Month | 1.7 (2.7) | 1.5 (2.1) | 0 (0)
  3 Months | .8 (1.6) | 0 (0) | 0 (0)
  6 Months | 0 (0) | 0 (0) | 0 (0)
  12 Months | 0 (0) | 0 (0) | 0 (0)

2. Secondary Outcome: Pain Score, Acute
Description: Acute Pain on Day 1, as measured by the Pain Quality Assessment Scale (PQAS). The scale goes from 0 (no pain) to 10 (the most intense pain sensation imaginable). Higher scores means worse pain.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BALANCED INHALATIONAL | TIVA-K | TIVA-R
Number analyzed (Participants) | 6 | 2 | 2
score on a scale | 4.6 (3.5) | 9.0 (0) | 3.0 (1.4)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | BALANCED INHALATIONAL | TIVA-K | TIVA-R
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT02527083/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT02527083/ICF_001.pdf